CLINICAL TRIAL: NCT04557332
Title: mHealth for ART Adherence by HIV+ African Americans Age 45 & Older
Brief Title: mHealth for ART Adherence by HIV+ African Americans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Collaborators: Prisma Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R44MD007161-05 (NIH)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which participants were randomly assigned to intervention group or control group.
Who Masked: Outcomes Assessor
Masking Description: Investigators and participants were aware of which group participants were randomly assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app (Experimental): In this arm, participants received a mobile app to support ART medication adherence.
  Interventions: Behavioral: On the Dot Mobile app
- Control (No Intervention): In this arm, participants received care as usual.

INTERVENTIONS:
Behavioral: On the Dot Mobile app — On the Dot is a mobile app to support HIV medication adherence. The mobile app is linked to a clinician portal through which participants can receive adherence support.
  Arms: Mobile app

SUMMARY:
The objective of this grant is to create and test a mobile app to support ART adherence among HIV+ African American adults.

DETAILED DESCRIPTION:
The Phase II project will enhance the existing (Phase 1) mobile intervention by offering: 1) a two-way communication capability through which participants can: i) indicate "pill taken" in response to pill reminders, and ii) receive a positive visual icon as behavioral-economics based reinforcement for "pill taken" responses; 2) pharmacist counseling and medication support; and, 3) the addition of educational and motivational text messages. Overall aims are to: 1) expand mhealth intervention to incorporate new Phase II features; 2) evaluate effectiveness in an RCT of HIV+ African Americans; and 3) prepare marketing and commercialization plans. Our long-term goal is to increase ART medication adherence, thus decreasing health disparities, among HIV+, African-Americans.

ELIGIBILITY:
Inclusion Criteria:

(a) self-identify as African American, (b) age 30 or older, (c) HIV positive (d) currently on ART (e) report having problems with, and interest in improving their ART adherence (f) own a smartphone (g) report English as their primary language

-

Exclusion Criteria:

(a) not self-identified as African American, (b) under age 30 (c) HIV negative (d) not currently on ART (e) do not report having problems with, or interest in, improving their ART adherence (f) do not own a smartphone (g) do not report English as a primary language and (h) participating in another research study or clinical trial (i) receiving care at non-participating site and, (j) dementia diagnosis.

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Self-reported ART medication adherence | 90 days
  Adherence was assessed using a 3-item self-report measure examining ART use in the prior 7 days, a time period, which is considered a reliable indictor of overall adherence (Bianco et al., 2010; Kleeburger et al., 2001; Segeral et al., 2010; Spire et al. 2008). The measure consists of a yes or no response to each of the following three questions: (i) "did you miss any ART doses during the last four days?," (ii) "Were you late for any of your intakes by more than two hours during the last four days?," and (iii) "did you miss any ART doses last week-end?"

SECONDARY OUTCOMES:
HIV medication adherence self efficacy | 90 days
  HIV treatment self-efficacy was assessed using the 17-item self-efficacy belief subscale of the modified HIV Medication Taking Self-Efficacy Scale.
Stress Burden | 90 days
  Stress burden will be assessed using the Perceived Stress Scale (Cohen et al., 1983), a well-validated instrument used with diverse populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No